CLINICAL TRIAL: NCT02597842
Title: Efficiency of Transcutaneous Electrical Acupoint Stimulation(TEAS) With Single Acupoint or Two Acupoints for Postoperative Nausea and Vomiting in Laparoscopic Operation: A Single Center, Randomized, Double-blinded, Controlled Clinical Trial
Brief Title: Transcutaneous Electrical Acupoint Stimulation(TEAS) for Postoperative Nausea and Vomiting in Laparoscopic Operation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: wangqiang (Other)
Responsible Party: Sponsor-Investigator, wangqiang, Professor, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: xijingmazui79
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative nausea and vomiting; TEAS
MeSH Terms: conditions — Postoperative Nausea and Vomiting

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- shuangxuezu (Experimental): Patients were given 30min of TEAS before induction until the end of the operation at two acupoints.
  Interventions: Device: TEAS (transcutaneous electrical acupoint stimulation)
- neiguanxuezu (Experimental): Patients were given TEAS at neiguan acupoint.
  Interventions: Device: TEAS (transcutaneous electrical acupoint stimulation)
- zusanlixuezu (Experimental): Patients were given TEAS at Zusanli acupoint.
  Interventions: Device: TEAS (transcutaneous electrical acupoint stimulation)
- duizhaozu (Sham Comparator): Patients were not given TEAS at two acupoints.
  Interventions: Device: TEAS (transcutaneous electrical acupoint stimulation)

INTERVENTIONS:
Device: TEAS (transcutaneous electrical acupoint stimulation) — Electric stimulation was given through electrode attached to specific acupoints

SUMMARY:
This is a single center, randomized, double-blinded, controlled clinical trial.The purpose of this study is to compare the effect of TEAS pretreatment with single acupoint or two acupoints for postoperative nausea and vomiting in patients undergoing laparoscopic operation.

DETAILED DESCRIPTION:
Patients were randomly assigned to four groups, receiving TEAS 30 minutes before induction.The stimulation was applied until the end of the operation. Postoperative nausea and vomiting was recorded 30 minute, 2 hour, 6 hour and 24 hour after the operation. The adverse events were recorded as well.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I-III
2. Aged 18 to 65 years old
3. Scheduled for general anesthesia
4. BMI index is between 18 to 30
5. Informed consented

Exclusion Criteria:

1. ASA IV
2. Hypertension that is not controlled
3. Severe hepatic or renal dysfunction
4. Ever had received electrical stimulation treatment
5. Severe systemic infection
6. With contraindications to the use of TEAS, such as skin damage or infection at the acupoints
7. For any reason one can not cope with the studies, such as the following:

   language comprehension, mental illness
8. Participate in the other clinical trial 3 month before the enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-08 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative nausea and vomiting | within 24 hours after operation

SECONDARY OUTCOMES:
Incidence of other postoperative complications | 30minutes, 2hours, 6hours and 24 hours after operation
Postoperative nausea and vomiting（PONV） score | 30minutes, 2hours, 6hours and 24 hours after operation
Visual Analogue Scale (VAS) pain score in PACU | 30 minutes after operation
Change of concentration of serum 5-HT | intraoperative
Change of concentration of serum dopamine | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Lizhe Xiong, M.D.;Ph D, Study Chair — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi, China